CLINICAL TRIAL: NCT03010449
Title: A Single Arm Pilot Study of Lung Volume Reduction in Severe Emphysema Using Bronchoscopic Autologous Blood Instillation in Combination With Intra-bronchial Valves
Brief Title: LVR in Severe Emphysema Using Bronchoscopic Autologous Blood Instillation in Combination With Intra-bronchial Valves
Acronym: BLOOD-VALVES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 135459
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema
Keywords: Lung volume reduction treatment; Autologous blood instillation; Intra-bronchial valve (IBV); Endobronchial valve
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-bronchial valve and blood (Experimental): Bronchoscopic lung volume reduction using intra-bronchial valves combined with autologous blood instillation.
  Interventions: Device: Intra-bronchial valve and blood

INTERVENTIONS:
Device: Intra-bronchial valve and blood — Intra-bronchial valve implantation in combination with autologous blood instillation

SUMMARY:
A single arm pilot study of lung volume reduction in severe emphysema using bronchoscopic autologous blood instillation in combination with intra-bronchial valves.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is an umbrella term encompassing two entities causing progressive and ultimately disabling breathlessness. Emphysema is a process destructive of the airspaces distal to the terminal bronchioles, with loss of gas exchange tissue, of elastic recoil and of circumferential tethering of the small airways leading to their collapse on forced expiration. Chronic bronchitis is a disorder of the bronchi causing excess production and impaired mobilisation of mucus. Increased parasympathetic tone and progressive remodelling of airways impairs response to bronchodilators. Static and dynamic hyperinflation with a persistently expanded chest and flattened diaphragms despite increasing use of accessory respiratory muscles results in a disadvantaged respiratory pump.

Patients with severe emphysema and hyperinflation may benefit from lung volume reduction techniques designed to reduce gas trapping and to improve airflow, chest wall and lung mechanics. The best evidence exists for lung volume reduction surgery (LVRS), which however is not without risk and there is increasing interest in the development of bronchoscopic lung volume reduction (BLVR) techniques including emplacement of intra-bronchial valves and bronchoscopic instillation of blood products, which have been shown individually to improve lung function, exercise capacity, and quality of life.

Most of the experience in bronchoscopic lung volume reduction has been with endobronchial valves which were introduced in 2001. One-way valves are inserted into segmental airways to deflate the most emphysematous lobes of the lung, allowing compromised lesser diseased tissue to expand and regain its function. Reduction of hyperinflation and improved lung function, exercise capacity, and quality of life, have been observed using the intra-bronchial valve (IBV Valve System) by Olympus in patients with upper lobe-predominant emphysema. These improvements are most pronounced in those with radiologically intact lobar fissures, a surrogate observation thought to indicate an absence of collateral ventilation, which can be confirmed using the Chartis balloon catheter system. A combined approach of CT fissure analysis and Chartis measurement is suggested to ensure the appropriate selection of patients.

Bronchoscopic instillation of biological agents such as fibrinogen, thrombin or autologous blood into the sub-segmental airways induces lung volume reduction initially by airway obstruction and resorption atelectasis followed by a localised inflammatory reaction leading to tissue remodelling at the alveolar level, with fibrosis and contraction of the target lobe. Unlike the intra-bronchial valve, collateral ventilation is not an issue, seeming not to influence the outcome. The cost compares favourably with that of prosthetic implants. Preliminary data from phase 1 and 2 trials using fibrinogen and thrombin in patients with upper lobe-predominant emphysema demonstrated improvements in lung function, exercise capacity, and quality of life scores up to 6 months with a trend towards better outcomes in those receiving 20mls (versus 10mls) to each of eight sub-segmental sites (four per upper lobe). Most patients experienced a self-limiting inflammatory reaction characterised by fever, malaise, shortness of breath, pleuritic chest pain and/or leucocytosis within 24 hours. 11 of 50 patients (22%) in phase 2 experienced a procedure-related COPD exacerbation comparable to other forms of endoscopic lung volume reduction. Similar physiological and symptomatic outcomes were observed in patients with homogeneous emphysema with 20mls (versus 10mls) per sub-segment instillation. Bakeer et al compared bronchoscopic lung volume reduction in patients with heterogeneous emphysema using autologous blood (n=7) with fibrin glue (n=8). At 12 weeks, statistically significant improvements in hyperinflation, lung function, exercise capacity (6MWT), and quality of life scores were observed in both groups. COPD exacerbations were fewer compared to earlier studies, which the authors suggest may be due to the use of a triple lumen balloon catheter protecting surrounding sub-segments from overspill and unintended inflammatory responses.

The prospect of broadening the eligibility for intra-bronchial valve implantation to include those with collateral ventilation treated with autologous blood is attractive and not yet studied.

Furthermore, the mechanisms of actions of intra-bronchial valves and of autologous blood instillation are not fully understood and may extend beyond lung volume reduction. In valve procedures where volume reduction has not been achieved, clinically meaningful improvements in quality of life independent of lung function have been described. Recruitment of compressed lung, restoration of elastic recoil and redirection of airflow are some of the postulated effects that are likely to involve the small airways. This may be investigated, for example, with multiple breath nitrogen washout (MBNW) which is a sensitive marker of small airways disease and can measure ventilation inhomogeneity, functional residual capacity and estimate trapped gas volumes. Impulse oscillometry (IOS) yields information on airway resistance and reactance (a measure of compliance) and distinguishes between large and small airway resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 or older
2. Diagnosis of severe COPD
3. Stopped smoking for at least 6 months prior to entering the study.
4. Completed a pulmonary rehabilitation program within 12 months prior to treatment and/or regularly performing maintenance respiratory rehabilitation if initial supervised therapy occurred more than 12 months prior to baseline testing.
5. Received Influenza vaccination consistent with local recommendations and/or policy.
6. Read, understood and signed the Informed Consent form.
7. Dyspnea scoring ≥2 on mMRC scale of 0-4.
8. FEV1%pred <45% and FEV1/FVC <60%.
9. TLC%pred >100% AND RV%pred >175%.
10. RV/TLC >55%
11. CT thorax must demonstrate heterogeneous emphysema and a disrupted interlobar fissure (75-90% intact) in the treatment lobe. Scans will be analysed using in-house software to calculate a heterogeneity score and percentage fissure integrity.
12. Chartis balloon catheter assessment confirms the presence of collateral ventilation in the target lobe.

Exclusion Criteria:

1. Patient unable to provide informed consent.
2. Subject has a history of recurrent clinically significant respiratory infections, defined as 3 or more hospitalizations for respiratory infection during the year prior to enrolment.
3. Subject has clinically significant bronchiectasis.
4. Alpha-1 AT deficiency.
5. Medical history of asthma.
6. Subject has co-morbidities that may significantly reduce ability to improve exercise capacity (e.g., severe arthritis, planned knee surgery) or baseline limitation on 6MWT is not due to dyspnoea.
7. Subject has evidence of other severe disease (such as, but not limited to, lung cancer or renal failure), which in the judgment of the investigator may compromise survival of the subject for the duration of the study.
8. Subject is pregnant or lactating, or plans to become pregnant within the study timeframe.
9. Subject has an inability to tolerate bronchoscopy under conscious sedation or general anaesthesia.
10. Subject has severe gas exchange abnormalities as defined by: PaCO2 >8.0 kPa and/or PaO2 < 6.0 kPa (on room air).
11. FEV1 <15% predicted and Total lung CO uptake (TLCO) <20% predicted.
12. Subject has an inability to walk >140 meters in 6 minutes.
13. Subject has severe pulmonary hypertension defined by right ventricular systolic pressure >45 mm Hg measured on transthoracic echocardiogram.
14. Subject has giant bullae >1/3 lung volume.
15. Lung nodule requiring surgery.
16. Subject has had previous LVR surgery, lung transplantation or lobectomy.
17. Subject has been involved in pulmonary drug or device studies within 30 days prior to this study.
18. Subject is taking >10 mg prednisone (or equivalent dose of a similar steroid) daily.
19. Subject requires high level chronic immunomodulatory therapy to treat a moderate to severe chronic inflammatory autoimmune disorder.
20. Subject is on an antiplatelet (such as Plavix) or anticoagulant therapy (such as Warfarin or NOAC) which cannot be stopped prior to the procedure.
21. Subject has a known sensitivity or allergy to Nickel.
22. Subject has a known sensitivity to drugs required to perform bronchoscopy.
23. Subject has any other disease, condition(s) or habit(s) that would interfere with completion of study and follow up assessments, would increase risks of bronchoscopy or assessments, or in the judgment of the investigator would potentially interfere.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-24 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Change in FEV1 between baseline and 6 months follow-up after lung volume reduction treatment. | 6 months

SECONDARY OUTCOMES:
Change from baseline in CT lobar volumes 6 months post treatment | 6 months
Change from baseline in SGRQ 6 months post treatment | 6 months
Change from baseline in dyspnoea score 6 months post treatment | 6 months
Change from baseline in RV 6 months post treatment | 6 months
Change from baseline in TLC 6 months post treatment | 6 months
Change from baseline in RV/TLC 6 months post treatment | 6 months
Change from baseline in TLCO 6 months post treatment | 6 months
Change from baseline in lung compliance 6 months post-treatment | 6 months
Change from baseline in ventilation inhomogeneity 6 months post-treatment. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pallav L Shah, MBBS MD FRCP, Principal Investigator — Royal Brompton & Harefields Hospital
Locations (1):
- Royal Brompton & Harefields Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coxson HO, Nasute Fauerbach PV, Storness-Bliss C, Muller NL, Cogswell S, Dillard DH, Finger CL, Springmeyer SC. Computed tomography assessment of lung volume changes after bronchial valve treatment. Eur Respir J. 2008 Dec;32(6):1443-50. doi: 10.1183/09031936.00056008. Epub 2008 Aug 6. PMID 18684848
- [Result] Springmeyer SC, Bolliger CT, Waddell TK, Gonzalez X, Wood DE; IBV Valve Pilot Trials Research Teams. Treatment of heterogeneous emphysema using the spiration IBV valves. Thorac Surg Clin. 2009 May;19(2):247-53, ix-x. doi: 10.1016/j.thorsurg.2009.02.005. PMID 19662968
- [Result] Sterman DH, Mehta AC, Wood DE, Mathur PN, McKenna RJ Jr, Ost DE, Truwit JD, Diaz P, Wahidi MM, Cerfolio R, Maxfield R, Musani AI, Gildea T, Sheski F, Machuzak M, Haas AR, Gonzalez HX, Springmeyer SC; IBV Valve US Pilot Trial Research Team. A multicenter pilot study of a bronchial valve for the treatment of severe emphysema. Respiration. 2010;79(3):222-33. doi: 10.1159/000259318. Epub 2009 Nov 17. PMID 19923790
- [Result] Ninane V, Geltner C, Bezzi M, Foccoli P, Gottlieb J, Welte T, Seijo L, Zulueta JJ, Munavvar M, Rosell A, Lopez M, Jones PW, Coxson HO, Springmeyer SC, Gonzalez X. Multicentre European study for the treatment of advanced emphysema with bronchial valves. Eur Respir J. 2012 Jun;39(6):1319-25. doi: 10.1183/09031936.00019711. PMID 22654006
- [Result] Eberhardt R, Gompelmann D, Schuhmann M, Reinhardt H, Ernst A, Heussel CP, Herth FJF. Complete unilateral vs partial bilateral endoscopic lung volume reduction in patients with bilateral lung emphysema. Chest. 2012 Oct;142(4):900-908. doi: 10.1378/chest.11-2886. PMID 22459779
- [Result] Franke KJ, Nilius G, Domanski U, Ruhle KH. [Unilateral reduction of lung volume by application of intrabronchial valves on patients selected after endoscopic collateral ventilation assessment]. Pneumologie. 2014 Feb;68(2):100-5. doi: 10.1055/s-0033-1359025. Epub 2013 Dec 16. German. PMID 24343242
- [Result] Perch M, Riise GC, Hogarth K, Musani AI, Springmeyer SC, Gonzalez X, Iversen M. Endoscopic treatment of native lung hyperinflation using endobronchial valves in single-lung transplant patients: a multinational experience. Clin Respir J. 2015 Jan;9(1):104-10. doi: 10.1111/crj.12116. Epub 2014 Apr 15. PMID 24506317
- [Result] Wood DE, Nader DA, Springmeyer SC, Elstad MR, Coxson HO, Chan A, Rai NS, Mularski RA, Cooper CB, Wise RA, Jones PW, Mehta AC, Gonzalez X, Sterman DH; IBV Valve Trial Research Team. The IBV Valve trial: a multicenter, randomized, double-blind trial of endobronchial therapy for severe emphysema. J Bronchology Interv Pulmonol. 2014 Oct;21(4):288-97. doi: 10.1097/LBR.0000000000000110. PMID 25321447
- [Result] Szlubowska S, Zalewska-Puchala J, Majda A, Kocon P, Soja J, Gnass M, Pasko E, Cmiel A, Szlubowski A, Kuzdzal J. The influence of lung volume reduction with intrabronchial valves on the quality of life of patients with heterogeneous emphysema - a prospective study. Pneumonol Alergol Pol. 2015;83(6):418-23. doi: 10.5603/PiAP.2015.0069. PMID 26559793
- [Result] Snell GI, Holsworth L, Borrill ZL, Thomson KR, Kalff V, Smith JA, Williams TJ. The potential for bronchoscopic lung volume reduction using bronchial prostheses: a pilot study. Chest. 2003 Sep;124(3):1073-80. doi: 10.1378/chest.124.3.1073. PMID 12970040
- [Result] Toma TP, Hopkinson NS, Hillier J, Hansell DM, Morgan C, Goldstraw PG, Polkey MI, Geddes DM. Bronchoscopic volume reduction with valve implants in patients with severe emphysema. Lancet. 2003 Mar 15;361(9361):931-3. doi: 10.1016/S0140-6736(03)12762-6. PMID 12648974
- [Result] Koster TD, Slebos DJ. The fissure: interlobar collateral ventilation and implications for endoscopic therapy in emphysema. Int J Chron Obstruct Pulmon Dis. 2016 Apr 13;11:765-73. doi: 10.2147/COPD.S103807. eCollection 2016. PMID 27110109
- [Result] Ingenito EP, Reilly JJ, Mentzer SJ, Swanson SJ, Vin R, Keuhn H, Berger RL, Hoffman A. Bronchoscopic volume reduction: a safe and effective alternative to surgical therapy for emphysema. Am J Respir Crit Care Med. 2001 Jul 15;164(2):295-301. doi: 10.1164/ajrccm.164.2.2011085. PMID 11463604
- [Result] Ingenito EP, Berger RL, Henderson AC, Reilly JJ, Tsai L, Hoffman A. Bronchoscopic lung volume reduction using tissue engineering principles. Am J Respir Crit Care Med. 2003 Mar 1;167(5):771-8. doi: 10.1164/rccm.200208-842OC. Epub 2002 Oct 11. PMID 12406835
- [Result] Reilly J, Washko G, Pinto-Plata V, Velez E, Kenney L, Berger R, Celli B. Biological lung volume reduction: a new bronchoscopic therapy for advanced emphysema. Chest. 2007 Apr;131(4):1108-13. doi: 10.1378/chest.06-1754. PMID 17426216
- [Result] Criner GJ, Pinto-Plata V, Strange C, Dransfield M, Gotfried M, Leeds W, McLennan G, Refaely Y, Tewari S, Krasna M, Celli B. Biologic lung volume reduction in advanced upper lobe emphysema: phase 2 results. Am J Respir Crit Care Med. 2009 May 1;179(9):791-8. doi: 10.1164/rccm.200810-1639OC. Epub 2009 Jan 29. PMID 19179484
- [Result] Bakeer M, Abdelgawad TT, El-Metwaly R, El-Morsi A, El-Badrawy MK, El-Sharawy S. Low cost biological lung volume reduction therapy for advanced emphysema. Int J Chron Obstruct Pulmon Dis. 2016 Aug 3;11:1793-800. doi: 10.2147/COPD.S112009. eCollection 2016. PMID 27536091
- [Result] Refaely Y, Dransfield M, Kramer MR, Gotfried M, Leeds W, McLennan G, Tewari S, Krasna M, Criner GJ. Biologic lung volume reduction therapy for advanced homogeneous emphysema. Eur Respir J. 2010 Jul;36(1):20-7. doi: 10.1183/09031936.00106009. Epub 2009 Nov 19. PMID 19926742
- [Result] Lopes AJ, Mafort TT. Correlations between small airway function, ventilation distribution, and functional exercise capacity in COPD patients. Lung. 2014 Oct;192(5):653-9. doi: 10.1007/s00408-014-9626-1. Epub 2014 Jul 22. PMID 25047513